CLINICAL TRIAL: NCT04627428
Title: A Phase1/2a, Open-Label Study to Evaluate the Safety and Tolerability of RPE Stem Cell-derived RPE (RPESC-RPE) Transplantation as Therapy for Dry Age-related Macular Degeneration (AMD)
Brief Title: Safety and Tolerability of RPE Stem Cell-derived RPE(RPESC-RPE) Transplantation in Patients With Dry Age-related Macular Degeneration (AMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Luxa Biotechnology, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Regenerative Research Foundation (Unknown); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RPESC-RPE-01; U01EY030581 (NIH); UG3EY031810 (NIH)
Record Dates: First submitted 2020-11-01; First posted 2020-11-13 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 50,000 cells (Experimental): Six patients will receive single dose of 50,000 RPESC-RPE-4W cells in the eye.
  Interventions: Biological: RPESC-RPE-4W
- 150,000 cells (Experimental): Six patients will receive single dose of 150,000 RPESC-RPE-4W cells in the eye.
  Interventions: Biological: RPESC-RPE-4W
- 250,000 cells (Experimental): Six patients will receive single dose of 250,000 RPESC-RPE-4W cells in the eye.
  Interventions: Biological: RPESC-RPE-4W

INTERVENTIONS:
Biological: RPESC-RPE-4W — RPESC-RPE-4W

SUMMARY:
The main objective of the study is evaluation of the safety and tolerability of RPESC-RPE-4W as therapy for dry AMD.

DETAILED DESCRIPTION:
RPESC-RPE-4W is Allogeneic RPE stem cell (RPESC)-derived RPE cells (RPESC-RPE) isolated from the RPE layer of human cadaveric eyes are transplanted under the macular.

This first-in-human Phase 1/2a open-label dose-escalation interventional study plans to enroll a total of 18 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of dry AMD.
2. Ability to understand and give informed consent.
3. Adult male or female >55 years of age.
4. Medically suitable to undergo vitrectomy and subretinal injection (>60% on Karnofsky scale).
5. Postmenopausal if female (expected to be common for the age limitation), or the female partner of a male subject unable to father children.
6. If male, willing to use barrier and spermicidal contraception during the study.

Exclusion Criteria:

1. Allergy or hypersensitivity to dilation drops or fluorescein.
2. Active major medical conditions limiting ability to participate in the study.
3. Active malignancy or treatment with chemotherapy.
4. Systemic immunosuppressant therapy within past six months.
5. History of toxoplasmosis, retinal histoplasmosis or tuberculosis.
6. Receipt of investigational product (IP) in a clinical trial within prior six months.
7. Any other medical condition, which, in the Investigator's judgment, will interfere with the subject's ability to comply with the protocol, compromises subject safety, or interferes with the interpretation of the study results.
8. Pregnant or nursing females.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of RPESC-RPE-4W transplantation | 24 months
  The transplantation of RPESC-RPE-4W cells will be considered safe and tolerated in the absence of:
  * Decrease in visual acuity (VA) of more than 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (or to worse than counting fingers at three feet) from baseline
  * Any Grade 2 (CTCAE v5.0) or greater non-ocular Adverse Events (AE) related to the RPESC-RPE-4W investigational product (IP) or investigational interventions
  * Intraocular inflammation indicating contamination with an infectious agent or serious immune response greater than moderate severity related to the RPESC-RPE-4W investigational product or investigational interventions
  * Tumor formation > 1 mm size related to the IP or investigational interventions

SECONDARY OUTCOMES:
Change in the mean of Best Corrected Visual Acuity (BCVA) | 24 months
  Change in visual acuity will be measured by ETDRS chart.
Loss of ≥10 decibels of ten-degree average visual sensitivity microperimetry | 24 months
  Loss of ≥10 decibels of ten-degree average visual sensitivity will by measured by microperimetry.
Change in GA lesion area | 24 months
  Change in GA lesion area will be measured.
Evidence of structural changes | 24 months
  Structural evidence will be measured by OCT imaging, autofluorescence, fluorescein angiography, and fundus photography

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh C Rao, M.D., Principal Investigator — University of Michigan Kellogg Eye Center; Theodore Leng, MD, FACS, Principal Investigator — Spencer Center for Vision Research at Stanford University; David S Liao, MD, PhD, Principal Investigator — Retina-Vitreous Associates Medical Group
Locations (3):
- United States (3):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Spencer Center for Vision Research, Palo Alto, California
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No